CLINICAL TRIAL: NCT00475280
Title: "Geriatric Assessment Adapted" Therapy for Ph- ALL Elderly Patients. GIMEMA Protocol LAL1104. EudraCT Code 2005-002156-17
Brief Title: "Geriatric Assessment Adapted" Therapy for Ph- ALL Elderly Patients
Acronym: LAL1104
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL1104
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Leukemia, Lymphoblastic, Acute
Keywords: geriatric assessment adapted therapy; Leukemia, Lymphoblastic, Acute; Older patients; > 60 years old; Ph negative
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Geriatric assessment (Other)
  Interventions: Procedure: Geriatric assessment adapted therapy; Procedure: Stem cells autotransplantation

INTERVENTIONS:
Procedure: Geriatric assessment adapted therapy — Geriatric assessment is performed before the induction phase starts.
Procedure: Stem cells autotransplantation — Stem cells autotransplantation is performed after consolidation treatment

SUMMARY:
This study aims at considering clinical heterogeneity of patients based on a "geriatric assessment" without taking into account the real age of the subject. This will allow physicians to adapt therapy according to three different groups of patients: frail, fit and intermediate and to evaluate the efficacy and feasibility of a therapy adapted to the different categories of patients.

DETAILED DESCRIPTION:
Treatment:

1. Frail patients:

   * Pretreatment with PDN
   * Induction with Vinblastine and PDN
   * Maintenance with MTX, 6-MP, VBL and PDN
2. Fit patients:

   * Pretreatment with PDN
   * Induction with VCR, DNR and PDN
   * Consolidation with MTX, ARA-C and G-CSF
   * Autologous transplantation
   * Maintenance with MTX, 6-MP, VCR, and PDN
3. Intermediate patients:

   * Pretreatment with PDN
   * Induction with VCR, DNR and PDN
   * Consolidation with MTX, ARA-C and G-CSF
   * A second cycle of consolidation therapy
   * Maintenance with MTX, 6-MP, VCR, and PDN

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years old
* Cytomorphologic and immunophenotypic diagnosis of ALL (all FAB groups except L3 and all immunophenotypes except SmIg+ B-ALL)
* Signed informed consent

Exclusion Criteria:

* Age <= 60 years old
* Ph+ ALL
* Refuse to sign informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Overall survival in Ph negative ALL patients stratified according to a geriatric assessment | at 6 months from diagnosis for the Frail group of pts and at 2 years from diagnosis for the Fit and Intermediate group of patients

SECONDARY OUTCOMES:
Complete Response rate | After induction therapy
Stem cell autotransplant feasibility | At 6 months from diagnosis
Incidence of adult ALL | At diagnosis
Evaluation of molecular, cytogenetics and immunophenotype heterogeneity in ph negative ALL patients >60 | At diagnosis and during follow-up
Disease free survival | During follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felicetto FERRARA, Dr., Principal Investigator — Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli" di Napoli
Locations (32):
- Italy (32):
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Pagani, (SA)
  - Nuovo Ospedale "Torrete", Ancona
  - USL 8 - Ospedale S.Donato, Arezzo
  - Az. Ospedaliera S. G. Moscati, Avellino
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Marche U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Marche
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Ferrara
  - Divisione Ematologia 1 - Azienda Ospedaliera Universitaria "San Martino", Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Centro Oncologico Modenese - Dipartimento di Oncoematologia, Modena
  - Azienda Ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università Federico II, Napoli
  - Inferiore U.O. Medicina Interna Ematologia ed Oncologia P.O. Umberto I, Nocera Inferiore
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga, Orbassano
  - La Maddalena Casa di Cura di Alta Specialità Dipartimento Oncologico di III Livello, Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - UO di Ematologia Centro Oncologico Basilicata, Rionero in Vulture
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Segreteria di Ematologia - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - U.O. di Oncoematologia -plesso ospedaliero "A. Tortora" di Pagani, Salerno
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Clinica Ematologica - Policlinico Universitario, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandler DP, Ross JA. Epidemiology of acute leukemia in children and adults. Semin Oncol. 1997 Feb;24(1):3-16. PMID 9045302
- [Background] Taylor PR, Reid MM, Bown N, Hamilton PJ, Proctor SJ. Acute lymphoblastic leukemia in patients aged 60 years and over: a population-based study of incidence and outcome. Blood. 1992 Oct 1;80(7):1813-7. PMID 1382705
- [Background] Taylor PR, Reid MM, Proctor SJ. Acute lymphoblastic leukaemia in the elderly. Leuk Lymphoma. 1994 May;13(5-6):373-80. doi: 10.3109/10428199409049625. PMID 8069181
- [Background] Kantarjian HM, O'Brien S, Smith T, Estey EH, Beran M, Preti A, Pierce S, Keating MJ. Acute lymphocytic leukaemia in the elderly: characteristics and outcome with the vincristine-adriamycin-dexamethasone (VAD) regimen. Br J Haematol. 1994 Sep;88(1):94-100. doi: 10.1111/j.1365-2141.1994.tb04982.x. PMID 7803263
- [Background] Delannoy A, Ferrant A, Bosly A, Chatelain C, Doyen C, Martiat P, Michaux JL, Sokal G. Acute lymphoblastic leukemia in the elderly. Eur J Haematol. 1990 Aug;45(2):90-3. doi: 10.1111/j.1600-0609.1990.tb00424.x. PMID 2209825
- [Background] Spath-Schwalbe E, Heil G, Heimpel H. Acute lymphoblastic leukemia in patients over 59 years of age. Experience in a single center over a 10-year period. Ann Hematol. 1994 Dec;69(6):291-6. doi: 10.1007/BF01696557. PMID 7993936
- [Background] Ferrari A, Annino L, Crescenzi S, Romani C, Mandelli F. Acute lymphoblastic leukemia in the elderly: results of two different treatment approaches in 49 patients during a 25-year period. Leukemia. 1995 Oct;9(10):1643-7. PMID 7564503
- [Background] Bassan R, Di Bona E, Lerede T, Pogliani E, Rossi G, D'Emilio A, Buelli M, Rambaldi A, Viero P, Rodeghiero F, Barbui T. Age-adapted moderate-dose induction and flexible outpatient postremission therapy for elderly patients with acute lymphoblastic leukemia. Leuk Lymphoma. 1996 Jul;22(3-4):295-301. doi: 10.3109/10428199609051761. PMID 8819079
- [Background] Delannoy A, Sebban C, Cony-Makhoul P, Cazin B, Cordonnier C, Bouabdallah R, Cahn JY, Dreyfus F, Sadoun A, Vernant JP, Gay C, Broustet A, Michaux JL, Fiere D. Age-adapted induction treatment of acute lymphoblastic leukemia in the elderly and assessment of maintenance with interferon combined with chemotherapy. A multicentric prospective study in forty patients. French Group for Treatment of Adult Acute Lymphoblastic Leukemia. Leukemia. 1997 Sep;11(9):1429-34. doi: 10.1038/sj.leu.2400780. PMID 9305593
- [Derived] Piciocchi A, Messina M, Elia L, Vitale A, Soddu S, Testi AM, Chiaretti S, Mancini M, Albano F, Spadano A, Krampera M, Bonifacio M, Cairoli R, Vetro C, Colella F, Ferrara F, Cimino G, Bassan R, Fazi P, Vignetti M. Prognostic impact of KMT2A-AFF1-positivity in 926 BCR-ABL1-negative B-lineage acute lymphoblastic leukemia patients treated in GIMEMA clinical trials since 1996. Am J Hematol. 2021 Sep 1;96(9):E334-E338. doi: 10.1002/ajh.26253. Epub 2021 Jun 9. No abstract available. PMID 34048072
- See also: GIMEMA's Web page — http://www.gimema.it